CLINICAL TRIAL: NCT01926457
Title: Treating Prediabetes in the First Trimester: A Randomized Controlled Trial
Brief Title: Treating Prediabetes in the First Trimester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); Society for Maternal-Fetal Medicine (Unknown)
Responsible Party: Principal Investigator, Hilary Roeder, MD, Physican, Clinical Instructor, Maternal-Fetal Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSD-GDM-RCT
Record Dates: First submitted 2013-08-15; First posted 2013-08-21 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Prediabetes; Gestational Diabetes
Keywords: First trimester treatment of prediabetes; First trimester treatment of gestational diabetes; Umbilical cord C-Peptide; Neonatal fat mass; Gestational weight gain; Infant obesity
MeSH Terms: conditions — Prediabetic State; Diabetes, Gestational; Gestational Weight Gain; Pediatric Obesity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First Trimester Treatment of Prediabetes (Experimental): Patients randomized to first trimester treatment will receive the following intervention immediately initiated upon diagnosis of prediabetes at <15 weeks 0 days gestation
  * diabetes education
  * blood glucose monitoring
  * medications as needed per California Diabetes and Pregnancy established protocol
  * growth ultrasounds
  * antenatal testing
  Interventions: Other: Treatment of Prediabetes
- Third Trimester Treatment of Prediabetes (Active Comparator): Patients randomized to third trimester treatment will receive the following intervention to be initiated at 28 weeks of gestation
  * diabetes education
  * blood glucose monitoring
  * medications as needed per California Diabetes and Pregnancy established protocol
  * growth ultrasounds
  * antenatal testing
  Interventions: Other: Treatment of Prediabetes

INTERVENTIONS:
Other: Treatment of Prediabetes — Standardized treatment of prediabetes per California Diabetes and Pregnancy Program "Sweet Success"
  * diabetes education
  * blood glucose monitoring
  * medications as needed per California Diabetes and Pregnancy established protocol
  * growth ultrasounds
  * antenatal testing

SUMMARY:
The investigators plan to study a sample of women with prediabetes (diagnosed by Hemoglobin A1c (HbA1c) 5.7-6.4% or fasting plasma glucose (FPG) 92-125 mg/dL) in the first trimester of pregnancy, and patients will be randomized to first trimester or third trimester treatment; the first trimester group will receive intervention immediately upon diagnosis of prediabetes whereas the third trimester group will receive only routine prenatal care until 28 weeks at which time they will receive intervention.

Intervention is defined as:

* diabetes education
* blood glucose monitoring
* medications as needed
* growth ultrasounds
* antenatal testing

The primary outcome is umbilical cord C-Peptide >90th percentile. Secondary outcomes include neonatal fat mass at delivery, infant weight-for-length at 12 months of age, maternal gestational weight gain, and biomarkers (chemicals) measured in the placenta and the baby's umbilical cord blood.

The investigators hypothesize that women who undergo the above intervention in the first trimester will deliver significantly fewer neonates with umbilical cord C-Peptide >90th percentile, and that the neonates will have lower fat mass, and weight-for-length at 12 months. The investigators further hypothesize that a greater proportion of patients undergoing first trimester intervention will have appropriate maternal gestational weight gain as defined by the Institute of Medicine, and a greater proportion will return to prepregnancy weight within 12 months.

DETAILED DESCRIPTION:
The primary aim of the proposed research is to demonstrate that promoting a normoglycemic intrauterine milieu in women with prediabetes diagnosed in the first trimester of pregnancy with a Hemoglobin A1c (HbA1c) 5.7-6.4% or fasting plasma glucose (FPG) 92-125 mg/dL will decrease the accumulation of fetal white adipose tissue and development of infant/child obesity during the first year of life. This project is built upon the hypothesis that pregnant subjects with prediabetes randomized in the first trimester of pregnancy to strict glycemic control and pharmacotherapy as needed will have less fetal adiposity and adverse neonatal outcomes than those who receive the diagnosis of prediabetes but do not initiate care until the third trimester.

In the proposed study, 240 women meeting the above criteria for prediabetes at ≤ 15w0d gestation will be randomized to either first trimester or third trimester treatment. Each group will have diabetes education, initiate blood glucose monitoring, begin pharmacotherapy as needed (per established protocol), undergo growth ultrasounds, and antenatal testing. The first trimester arm will receive the above interventions immediately upon diagnosis of prediabetes whereas the third trimester arm will receive only routine prenatal care until 28 weeks at which time they will begin education and treatment. Both groups will be treated identically from 28 weeks until delivery.

In the 2013 the National Institutes of Health (NIH) Gestational Diabetes (GDM) Consensus Conference, the panel was concerned about adopting criteria that would increase prevalence of GDM (i.e. first trimester treatment) without first demonstrating improved outcomes. The results of this proposed trial, will allow us to fill key research gaps; this is the first prospective trial to evaluate the International Associations of Diabetes in Pregnancy Study Groups (IADPSG) recommendations for screening and diagnosing prediabetes in the first trimester.

Findings from this research will quantify the maternal and neonatal benefits and harms of treating women with prediabetes from early pregnancy. Additionally, the cohort of neonates that will result from this study can be followed into childhood to evaluate whether first trimester treatment has benefits beyond those anticipated at birth and may decrease the long-term incidence of obesity and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 and above
* Any ethnic background
* English- or Spanish-speaking
* Planned prenatal care/delivery at The University of California, San Diego's Hillcrest Hospital
* Singleton pregnancy
* Prediabetes diagnosed prior to 15w0d with HbA1c 5.7-6.4% or FPG 92-125 mg/dL

Exclusion Criteria:

* Known Type 2 Diabetes (T2DM)
* T2DM diagnosed with first trimester screening
* Patients with known maternal/fetal indications for delivery <36w0d
* Patients presenting for care after 15w0d

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Umbilical Cord C-Peptide >90th percentile | 1 day (Collected at the time of delivery)

SECONDARY OUTCOMES:
Neonatal fat mass | Within 48 hours of delivery
  Neonatal fat mass will be measured using an anthropometric model using weight, length, and flank skinfold thickness.
Adherence to the Institute of Medicine (IOM) guidelines for gestational weight gain | Weight gain will be measured from immediately preconception until delivery
  The IOM recommends that underweight women (BMI<18.5kg/m2) gain 28-40lbs, normal women (BMI 18.5-24.9 kg/m2) gain 25-35lbs, overweight women (BMI 25.0-29.9 kg/m2) gain 15-25lbs and obese women (BMI≥30 kg/m2) gain 11-20 lbs.
Return to prepregnancy weight | After 1 year post delivery

OTHER OUTCOMES:
birthweight | At delivery
birthweight percentile | At delivery
Infant gender | At delivery
Ponderal index | At delivery
  Weight/length^3
Neonatal Intensive Care Unit (NICU) Admission | Within 10 days after birth
Infant weight-for-length | 6 months and 12 months after delivery
Need for pharmacotherapy to control hyperglycemia | From 5 weeks gestation until time of delivery
Birth trauma | At delivery
  Shoulder dystocia, brachial plexus injury
Mode of delivery | At delivery
  Spontaneous delivery, operative vaginal delivery, cesarean delivery
Indication for delivery | At delivery
Total gestational weight gain | From immediately preconception until delivery
Postpartum weight retention | Within 1 year of delivery
Diagnosis of Preeclampsia | From 20 weeks gestation until 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Hilary A Roeder, MD, Principal Investigator — UC San Diego Health System; Gladys A Ramos, MD, Principal Investigator — UC San Diego Health System; Thomas R Moore, MD, Principal Investigator — UC San Diego Health System
Locations (1):
- UC San Diego Health System, San Diego, California, United States

REFERENCES:
- [Background] HAPO Study Cooperative Research Group. Hyperglycemia and Adverse Pregnancy Outcome (HAPO) Study: associations with neonatal anthropometrics. Diabetes. 2009 Feb;58(2):453-9. doi: 10.2337/db08-1112. Epub 2008 Nov 14. PMID 19011170
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Catalano PM, Thomas A, Huston-Presley L, Amini SB. Increased fetal adiposity: a very sensitive marker of abnormal in utero development. Am J Obstet Gynecol. 2003 Dec;189(6):1698-704. doi: 10.1016/s0002-9378(03)00828-7. PMID 14710101
- [Background] Kim SY, Sharma AJ, Callaghan WM. Gestational diabetes and childhood obesity: what is the link? Curr Opin Obstet Gynecol. 2012 Dec;24(6):376-81. doi: 10.1097/GCO.0b013e328359f0f4. PMID 23000698
- [Background] Catalano PM, McIntyre HD, Cruickshank JK, McCance DR, Dyer AR, Metzger BE, Lowe LP, Trimble ER, Coustan DR, Hadden DR, Persson B, Hod M, Oats JJ; HAPO Study Cooperative Research Group. The hyperglycemia and adverse pregnancy outcome study: associations of GDM and obesity with pregnancy outcomes. Diabetes Care. 2012 Apr;35(4):780-6. doi: 10.2337/dc11-1790. Epub 2012 Feb 22. PMID 22357187
- [Background] Hedderson MM, Gunderson EP, Ferrara A. Gestational weight gain and risk of gestational diabetes mellitus. Obstet Gynecol. 2010 Mar;115(3):597-604. doi: 10.1097/AOG.0b013e3181cfce4f. PMID 20177292
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Catalano PM, Thomas AJ, Avallone DA, Amini SB. Anthropometric estimation of neonatal body composition. Am J Obstet Gynecol. 1995 Oct;173(4):1176-81. doi: 10.1016/0002-9378(95)91348-3. PMID 7485315
- [Background] Riskin-Mashiah S, Younes G, Damti A, Auslender R. First-trimester fasting hyperglycemia and adverse pregnancy outcomes. Diabetes Care. 2009 Sep;32(9):1639-43. doi: 10.2337/dc09-0688. Epub 2009 Jun 23. PMID 19549728
- [Background] Persson B, Heding LG, Lunell NO, Pschera H, Stangenberg M, Wager J. Fetal beta cell function in diabetic pregnancy. Amniotic fluid concentrations of proinsulin, insulin, and C-peptide during the last trimester of pregnancy. Am J Obstet Gynecol. 1982 Oct 15;144(4):455-9. PMID 6751089
- [Background] Lappas M, Andrikopoulos S, Permezel M. Hypoxanthine-xanthine oxidase down-regulates GLUT1 transcription via SIRT1 resulting in decreased glucose uptake in human placenta. J Endocrinol. 2012 Apr;213(1):49-57. doi: 10.1530/JOE-11-0355. Epub 2012 Jan 19. PMID 22266962
- [Background] Gillum MP, Kotas ME, Erion DM, Kursawe R, Chatterjee P, Nead KT, Muise ES, Hsiao JJ, Frederick DW, Yonemitsu S, Banks AS, Qiang L, Bhanot S, Olefsky JM, Sears DD, Caprio S, Shulman GI. SirT1 regulates adipose tissue inflammation. Diabetes. 2011 Dec;60(12):3235-45. doi: 10.2337/db11-0616. PMID 22110092
- [Background] Banks AS, Kon N, Knight C, Matsumoto M, Gutierrez-Juarez R, Rossetti L, Gu W, Accili D. SirT1 gain of function increases energy efficiency and prevents diabetes in mice. Cell Metab. 2008 Oct;8(4):333-41. doi: 10.1016/j.cmet.2008.08.014. PMID 18840364
- [Background] Astapova O, Leff T. Adiponectin and PPARgamma: cooperative and interdependent actions of two key regulators of metabolism. Vitam Horm. 2012;90:143-62. doi: 10.1016/B978-0-12-398313-8.00006-3. PMID 23017715
- [Background] Qiao L, Yoo HS, Madon A, Kinney B, Hay WW Jr, Shao J. Adiponectin enhances mouse fetal fat deposition. Diabetes. 2012 Dec;61(12):3199-207. doi: 10.2337/db12-0055. Epub 2012 Aug 7. PMID 22872236
- [Background] Luo ZC, Nuyt AM, Delvin E, Fraser WD, Julien P, Audibert F, Girard I, Shatenstein B, Deal C, Grenier E, Garofalo C, Levy E. Maternal and fetal leptin, adiponectin levels and associations with fetal insulin sensitivity. Obesity (Silver Spring). 2013 Jan;21(1):210-6. doi: 10.1002/oby.20250. PMID 23505188
- See also: The American Association of Obstetricians and Gynecologists Foundation — http://www.aaogf.org/
- See also: UC San Diego Health System Department of Reproductive Medicine — http://repromed.ucsd.edu/